CLINICAL TRIAL: NCT03682952
Title: Evaluation of Nail Fold Microcirculation and Interventional Therapy in Patients With Chronic Renal Failure
Brief Title: Evaluation of Nail Fold Microcirculation in CKD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XYFY2018-KL034-01
Record Dates: First submitted 2018-09-12; First posted 2018-09-25 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-06

CONDITIONS: Chronic Renal Disease
Keywords: Chronic Renal Disease; Nail fold microcirculation; Interventional therapy
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Alprostadil; beraprost

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Alprostadil and Beraprost sodium tablets are used to improve the microcirculation of CKD patients.
  Interventions: Drug: Alprostadil Injection; Drug: Beraprost sodium tablets
- Anemia control group (No Intervention): Anemia patients
- Control group (No Intervention): Healthy person

INTERVENTIONS:
Drug: Alprostadil Injection — Participants are given alprostadil injection 10ug intravenously once a day for 2 weeks.
  Arms: Experimental group
Drug: Beraprost sodium tablets — Participants are given alprostadil injection 10ug intravenously once a day for 2 weeks ,then they take beraprost sodium tablets 40ug orally three times perday for 3 months.
  Arms: Experimental group

SUMMARY:
To evaluation of nailfold microcirculation in patients with chronic renal failure and its intervention therapy

DETAILED DESCRIPTION:
The aim of this study is to study the changes of Nailfold Microcirculation in patients with chronic renal failure, to clarify the correlation between the changes of Nailfold Microcirculation and renal function, and to explore whether nailfold microcirculation can be used as an indicator of renal microcirculation in patients with chronic renal failure, and to provide a noninvasive method for the clinical evaluation of renal microcirculation in patients with chronic renal failure.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients
* Without dialysis
* Blood pressure ≤ 140/90mmHg

Exclusion Criteria:

* Polycystic kidney
* Endocrine system disease
* Cardio-cerebrovascular disease
* Rheumatic immune disease
* Peripheral vascular disease
* Hematological diseases
* Respiratory disease
* Infection

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Nailfold microcirculation morphological integral | Up to three and a half months
  Nail fold capillary microscopy examination
Nailfold microcirculation blood flow integral | Up to three and a half months
  Nail fold capillary microscopy examination
Nail fold microcirculation perivascular loop integral | Up to three and a half months
  Nail fold capillary microscopy examination

SECONDARY OUTCOMES:
The content of blood serum creatinine | Up to three and a half months
  Intravenous blood sampling
The content of blood urea nitrogen | Up to three and a half months
  Intravenous blood sampling，uronoscopy
The content of blood cystatin C | Up to three and a half months
  Intravenous blood sampling
eGFR | Up to three and a half months
  Intravenous blood sampling
The content of blood albumin | Up to three and a half months
  Intravenous blood sampling
The quantification of urinary protein | Up to three and a half months
  Uronoscopy
The content of hemoglobin | Up to three and a half months
  Intravenous blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Dong Sun, MD, Study Director — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leunissen KM, van den Berg BW, Cheriex EC, Slaaf DW, Reneman RS, van Hooff JP. Influence of fluid removal during haemodialysis on macro- and skin microcirculation. Haemodynamic pathophysiologic study of fluid removal during haemodialysis. Nephron. 1990;54(2):162-8. doi: 10.1159/000185838. PMID 2314527
- [Background] Yuksel S, Pancar Yuksel E, Yenercag M, Soylu K, Zengin H, Gulel O, Meric M, Aydin F, Senturk N, Sahin M. Abnormal nail fold capillaroscopic findings in patients with coronary slow flow phenomenon. Int J Clin Exp Med. 2014 Apr 15;7(4):1052-8. eCollection 2014. PMID 24955181
- [Background] Senet P, Fichel F, Baudot N, Gaitz JP, Tribout L, Frances C. [Nail-fold capillaroscopy in dermatology]. Ann Dermatol Venereol. 2014 Jun-Jul;141(6-7):429-37. doi: 10.1016/j.annder.2014.04.120. Epub 2014 Jun 2. French. PMID 24951141
- [Background] Yuan SY. [Nail-fold microcirculatory flow in liver cirrhosis: diabetes mellitus and systemic lupus erythematosus]. Zhonghua Yi Xue Za Zhi. 1986 Aug;66(8):473-5, 512. No abstract available. Chinese. PMID 3096534
- [Background] Paparde A, Neringa-Martinsone K, Plakane L, Aivars JI. Nail fold capillary diameter changes in acute systemic hypoxia. Microvasc Res. 2014 May;93:30-3. doi: 10.1016/j.mvr.2014.02.013. Epub 2014 Mar 6. PMID 24607833
- [Background] Schumann L, Korten G, Holdt B, Holtz M. Microcirculation of the fingernail fold in CAPD patients: preliminary observations. Perit Dial Int. 1996 Jul-Aug;16(4):412-6. PMID 8863336
- [Background] Hasegawa K, Pereira BP, Pho RW. The microvasculature of the nail bed, nail matrix, and nail fold of a normal human fingertip. J Hand Surg Am. 2001 Mar;26(2):283-90. doi: 10.1053/jhsu.2001.21519. PMID 11279575